CLINICAL TRIAL: NCT00521430
Title: NON-T-CELL DEPLETED HLA-HAPLOIDENTICAL FAMILIAL DONOR HEMATOPOIETIC CELL TRANSPLANTATION AFTER REDUCED INTENSITY CONDITIONING
Brief Title: Donor Stem Cell Transplant After Conditioning Therapy in Treating Patients With Hematologic Cancer, Recurrent or Metastatic Solid Tumor, or Other Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000561542; AMC-UUCM-2004-0029
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2007-10

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Nonmalignant Neoplasm; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent childhood grade III lymphomatoid granulomatosis; childhood diffuse large cell lymphoma; recurrent childhood large cell lymphoma; childhood immunoblastic large cell lymphoma; recurrent childhood lymphoblastic lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; recurrent childhood small noncleaved cell lymphoma; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; aplastic anemia; recurrent childhood acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; refractory multiple myeloma; chronic myelomonocytic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; recurrent adult Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; adult nasal type extranodal NK/T-cell lymphoma; Waldenström macroglobulinemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; cutaneous B-cell non-Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; childhood chronic myelogenous leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; recurrent/refractory childhood Hodgkin lymphoma; secondary myelodysplastic syndromes; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Neoplasms; Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Extranodal NK-T-Cell; Burkitt Lymphoma; Anemia, Aplastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Waldenstrom Macroglobulinemia; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Recurrence | interventions — Antilymphocyte Serum; Busulfan; Cyclosporine; fludarabine phosphate; Methotrexate; Methylprednisolone; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: methotrexate
Drug: methylprednisolone
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor stem cell transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and methotrexate before and after transplant may stop this from happening.

PURPOSE: This clinical trial is studying the side effects and how well donor stem cell transplant works when given after conditioning therapy in treating patients with hematologic cancer, recurrent or metastatic solid tumor, or other disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of non-T-cell depleted, HLA-haploidentical related donor hematopoietic stem cell transplantation after a reduced-intensity conditioning regimen comprising busulfan, fludarabine phosphate, anti-thymocyte globulin, and methylprednisolone in patients with hematologic cancer, recurrent or metastatic solid tumors, or other diseases.

OUTLINE:

* Reduced-intensity conditioning regimen: Patients receive busulfan IV 4 times daily on days -7 and -6; fludarabine phosphate IV over 30 minutes on days -7 to -2; and methylprednisolone IV over 30 minutes followed by anti-thymocyte globulin IV over 4 hours on days -4 to -1.
* Donor hematopoietic stem cell transplantation: Patients receive donor peripheral blood stem cells IV over 1 hour on days 0 and 1.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV over 2-4 hours or orally twice daily beginning on day -1 and continuing until day 60, followed by a taper in the absence of GVHD. Patients also receive methotrexate IV on days 2, 4, 7, and 12.

After the transplant, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * High-risk acute leukemia, including any of the following:

    * Refractory acute leukemia
    * Acute leukemia beyond first remission
    * Acute leukemia in first remission with poor prognostic features (e.g., chromosomal changes suggesting poor prognosis)
  * Chronic myelogenous leukemia in second chronic, accelerated, or blastic phase
  * Severe aplastic anemia that is not responsive to immunosuppressive therapy
  * Myelodysplastic syndromes, including any of the following:

    * Refractory anemia (RA) or RA with ringed sideroblasts with severe cytopenia
    * RA with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia
  * Refractory or relapsed non-Hodgkin or Hodgkin lymphoma
  * Multiple myeloma
  * Biopsy proven measurable solid tumor meeting 1 of the following criteria:

    * Recurrent disease after primary treatment and deemed incurable to standard treatment
    * Metastatic disease for which no known standard therapy that is potentially curative or definitely capable of extending life expectancy exists
* Must have a related HLA-haploidentical mismatched (3/6 or fewer loci) donor available

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Bilirubin < 2.0 mg/dL
* AST < 3 times upper limit of normal
* Creatinine < 2.0 mg/dL
* Ejection fraction > 40% by MUGA

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-04; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Engraftment (neutrophil, platelet, and red blood cells)
Frequency and kinetics of mixed chimerism as assessed by polymerase chain reaction
Frequency and severity of regimen-related toxicities
Frequency of acute and chronic graft-versus-host disease
Immune reconstitution

SECONDARY OUTCOMES:
Tumor response rate
Duration of tumor response
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo H. Lee, MD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center - University of Ulsan College of Medicine, Seoul, South Korea

REFERENCES:
- [Result] Lee KH, Lee JH, Lee JH, Kim DY, Seol M, Lee YS, Kang YA, Jeon M, Hwang HJ, Jung AR, Kim SH, Yun SC, Shin HJ. Reduced-intensity conditioning therapy with busulfan, fludarabine, and antithymocyte globulin for HLA-haploidentical hematopoietic cell transplantation in acute leukemia and myelodysplastic syndrome. Blood. 2011 Sep 1;118(9):2609-17. doi: 10.1182/blood-2011-02-339838. Epub 2011 Jun 28. PMID 21715313